CLINICAL TRIAL: NCT02415660
Title: Short-Term Response of Thoracic Spine Manipulation With or Without Trigger Point Dry Needling for Mechanical Neck Pain: A Randomized Clinical Trial
Brief Title: Short-Term Response of Thoracic Spine Manipulation With or Without Trigger Point Dry Needling for Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Young, Assistant Professor, Army-Baylor Doctoral Program in PT, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 404153-1
Record Dates: First submitted 2015-03-25; First posted 2015-04-14 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Neck Pain
Keywords: trigger point dry needling; thoracic spine manipulation; deep cervical extensor muscle; deep cervical flexor muscle; shear wave elastography
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMT and TDN (Experimental): Thoracic spinal manipulation and trigger point dry needling using Seirin J-type stainless steel needles, 0-2-0.3 x 40-50 mm. Exercise program consists of cervical range of motion exercises and posterior neck muscle activation exercise.
  Interventions: Procedure: Thoracic spinal manipulation; Procedure: Trigger point dry needling; Behavioral: Cervical range of motion exercises; Behavioral: Posterior neck muscle activation exercise; Device: Seirin J-type stainless steel needles, 0-2-0.3 x 40-50 mm
- SMT and Sham TDN (Sham Comparator): Thoracic spinal manipulation and trigger point dry needling sham. Exercise program consists of cervical range of motion exercises and posterior neck muscle activation exercise.
  Interventions: Procedure: Thoracic spinal manipulation; Behavioral: Cervical range of motion exercises; Behavioral: Posterior neck muscle activation exercise; Procedure: Trigger point dry needling sham

INTERVENTIONS:
Procedure: Thoracic spinal manipulation — All patients will receive 3 different thrust joint manipulations to the middle and upper thoracic spine region. Each technique will be applied up to 2 times, per the discretion of the treating therapist discretion
Procedure: Trigger point dry needling — The TDN treatment will consist of a trained investigator inserting a needle through the participant's skin, into the deep cervical extensor muscles and/or the upper trapezius muscles using FDA approved (FDA regulation # 880.5580) disposable 0.2-0.3 x 40-50 mm stainless steel Seirin J-type needles (Seirin, Japan). Those subjects randomized to TDN will undergo this treatment.
  Arms: SMT and TDN
Behavioral: Cervical range of motion exercises — The patient will be instructed to place 5 fingers along the manubrium, and to flex the neck down until the chin touches the fingers. The patient will then be instructed to rotate the head as far as comfortably possible to one side, and then to the other side for 10 repetitions to each side, 3-4 times per day. The patient will progress from 5 fingers, to 4, 3, 2 and eventually 1 finger as neck mobility improves.
Behavioral: Posterior neck muscle activation exercise — The patient will be instructed to sit upright in a chair, and place 1-2 fingers over the C2 spinous process. Education to localize this landmark will be provided. The patient will then perform an isometric chin tuck exercise against the resistance they will apply at C2. This position will be held x 5 seconds and repeated 10 times, 3-4 times per day.
Procedure: Trigger point dry needling sham — The sham group will receive a simulated TDN. Using a toothpick in a needle guide-tube, the investigator will tap, rest, and twist the toothpick for approximately 30 seconds in the same 2 muscles, 2 sites in each muscle. The sham treatment will not penetrate the skin.
  Arms: SMT and Sham TDN
Device: Seirin J-type stainless steel needles, 0-2-0.3 x 40-50 mm — A trained investigator will insert the needle through the participants skin into the deep cervical extensors and/or the upper trapezius muscles. Needles are FDA approved (#880.5580)
  Arms: SMT and TDN

SUMMARY:
This study will assess the short term response of thoracic spinal manipulation with or without trigger point dry needling in 58 subjects with a primary complaint of mechanical neck pain.

DETAILED DESCRIPTION:
Neck pain is common, and return to duty rates after medical evacuation from theater for spinal pain is low. Muscles comprise the majority of the stability for the cervical spine, yet neck muscle function can be altered in the presence of pain. Research has consistently shown the benefit of including thoracic spine manipulation (SMT) in the treatment of patients with mechanical neck pain. Emerging evidence is now also showing promising benefit of including trigger point dry needling (TDN) for the treatment of mechanical neck pain. Treatment regimens commonly address anterior cervical stabilizing musculature, but little is known regarding the response to treatment of the deep posterior stabilizing musculature.

This study will assess the short term response of thoracic SMT with or without TDN in 58 subjects with a primary complaint of mechanical neck pain. Subjects will be randomized to receive 2 treatment visits approximately 2-3 days apart of either SMT+sham TDN or SMT+TDN. TDN will be directed to the upper trapezius and deep cervical extensor muscles of the neck. Outcomes of interest will be changes in function and pain. Assessments will be made at baseline, immediately after the first treatment, at the 2nd treatment, and approximately 5-7 days after the 2nd treatment visit. A subgroup of 20 subjects (10 per group) will also have the upper trapezius and deep cervical extensor muscle activation assessed via shear wave elastography, and deep cervical flexor activation assessed via the craniocervical flexion test.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64 years and eligible for military health care
2. Primary complaint of mechanical neck pain provoked by posture, movement or palpation of neck musculature, with or without unilateral upper extremity symptoms.
3. Presence of active trigger points in either the upper trapezius or deep cervical extensor muscles.
4. Able to make one initial appointment at the Army Medical Department Center and School at Fort Sam Houston, one treatment visit approximately 2-3 days after the initial visit, and then a final outcome visit approximately 5-7 days after 2nd visit.
5. No less than 10 points (0-50 range) on the Neck Disability Index.

Exclusion Criteria:

1. Prior history of whiplash injury resulting in neck pain which required medical treatment.
2. Any prior physical therapy, chiropractic, acupuncture treatment or injections for neck pain within the past 3 months.
3. History of cervical spine surgery.
4. History of any systemic disorder in which thoracic spine manipulation and TDN would be contraindicated (i.e. osteoporosis, bleeding disorders or anticoagulant medication use)
5. Signs and symptoms consistent with nerve root compression (i.e. diminished upper extremity strength, sensation or reflexes), cervical artery insufficiency (i.e. nystagmus, gait disturbances, Horner Syndrome) or upper cervical ligament instability (i.e. Sharp-Purser, alar ligament, transverse ligament tests).
6. Current primary complaint of headaches
7. Pending legal action regarding their neck pain
8. Inability to read and understand English
9. Females known or thought to be pregnant

   -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | Change in NDI from baseline to 2-3 days
  The NDI is a revised form of the Oswestry Low Back Pain Index. It is designed to measure the activities of daily living in persons with neck pain.
Change in Neck Disability Index (NDI) | Change in NDI at 7-10 days
  The NDI is a revised form of the Oswestry Low Back Pain Index. It is designed to measure the activities of daily living in persons with neck pain.

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) | Change in pain from baseline to 2-3 days
  An 11-point NPRS will be used to measure pain intensity. The scale is anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain".
Change in Numeric Pain Rating Scale (NPRS) | 7-10 days
  An 11-point NPRS will be used to measure pain intensity. The scale is anchored on the left with the phrase "No Pain" and on the right with the phrase "Worst Imaginable Pain".
Global Rate of Change (GRC) | 2-3 days
  The GRC assesses subjective perception of overall change over time and the importance of that change. A 15-point Likert type scale ranging from -7 (very great deal worse) to +7 (a very great deal better) will be used.
Global Rate of Change (GRC) | 7-10 days
  The GRC assesses subjective perception of overall change over time and the importance of that change. A 15-point Likert type scale ranging from -7 (very great deal worse) to +7 (a very great deal better) will be used.
Change in Deep cervical multifidus activation using ultrasound Shear Wave Elastography (SWE) | Day 1 pre and post intervention
  Shear-Wave Elastography (SWE) is an evolving technology that uses advanced ultrasound imaging to quantify tissue stiffness (i.e., elasticity). This technology will be utilized to assess change in passive muscle activation response to treatment.
Change in Deep cervical multifidus activation using ultrasound Shear Wave Elastography (SWE) | 7-10 days
  Shear-Wave Elastography (SWE) is an evolving technology that uses advanced ultrasound imaging to quantify tissue stiffness (i.e., elasticity). This technology will be utilized to assess change in passive muscle activation response to treatment.
Change in Deep Neck Flexor (DNF) Activation | Day 1 pre and post intervention
  Change in DNF muscle activation will be assessed via the chin tuck head lift test (CTHL).
Change in Deep Neck Flexor (DNF) Activation | 7-10 days
  Change in DNF muscle activation will be assessed via the chin tuck head lift test (CTHL).
Change in Pain Pressure Threshold (PPT) as assessed using an electronic algometer. | Day 1 pre and post intervention
  PPT is the minimal amount of pressure that produces pain and is used to assess abnormalities in nociceptive processing or hyperalgesia.
Change in Pain Pressure Threshold (PPT) as assessed using an electronic algometer. | 7-10 days
  PPT is the minimal amount of pressure that produces pain and is used to assess abnormalities in nociceptive processing or hyperalgesia.

CONTACTS AND LOCATIONS:
Overall Officials: David M Boland, PT, DPT, PhD, Principal Investigator — Assistant Professor, Army-Baylor Doctoral Program in PT
Locations (1):
- AMEDD Center & School, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker MJ, Boyles RE, Young BA, Strunce JB, Garber MB, Whitman JM, Deyle G, Wainner RS. The effectiveness of manual physical therapy and exercise for mechanical neck pain: a randomized clinical trial. Spine (Phila Pa 1976). 2008 Oct 15;33(22):2371-8. doi: 10.1097/BRS.0b013e318183391e. PMID 18923311
- [Background] O'Leary S, Cagnie B, Reeve A, Jull G, Elliott JM. Is there altered activity of the extensor muscles in chronic mechanical neck pain? A functional magnetic resonance imaging study. Arch Phys Med Rehabil. 2011 Jun;92(6):929-34. doi: 10.1016/j.apmr.2010.12.021. Epub 2011 May 6. PMID 21529779
- [Background] Schomacher J, Falla D. Function and structure of the deep cervical extensor muscles in patients with neck pain. Man Ther. 2013 Oct;18(5):360-6. doi: 10.1016/j.math.2013.05.009. Epub 2013 Jul 12. PMID 23849933
- [Background] Cleland JA, Mintken PE, Carpenter K, Fritz JM, Glynn P, Whitman J, Childs JD. Examination of a clinical prediction rule to identify patients with neck pain likely to benefit from thoracic spine thrust manipulation and a general cervical range of motion exercise: multi-center randomized clinical trial. Phys Ther. 2010 Sep;90(9):1239-50. doi: 10.2522/ptj.20100123. Epub 2010 Jul 15. PMID 20634268
- [Background] Maher RM, Hayes DM, Shinohara M. Quantification of dry needling and posture effects on myofascial trigger points using ultrasound shear-wave elastography. Arch Phys Med Rehabil. 2013 Nov;94(11):2146-50. doi: 10.1016/j.apmr.2013.04.021. Epub 2013 May 14. PMID 23684553